CLINICAL TRIAL: NCT06950957
Title: Comparison of Video Laryngeal Mask Airway and Endotracheal Tube Use for Airway Safety in Patients Undergoing Septoplasty
Brief Title: Video Laryngeal Mask vs. Endotracheal Tube in Septoplasty
Status: Recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKEAK 2025/3/15
Record Dates: First submitted 2025-03-24; First posted 2025-04-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Airway Complication of Anesthesia; Anesthesia Intubation Complication; Septoplasty
Keywords: Septoplasty; Laryngeal Mask Airway; Endotracheal Tube; Postoperative Sore Throat; Airway Leak; Otorhinolaryngology Surgery; Supraglottic Airway Devices; Aldrete Score; Postoperative Sore Throat (POST Score)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VLMA Group: Participants assigned to this group will receive airway management via a video laryngeal mask airway (VLMA) with an integrated camera system for direct visualization of the laryngeal inlet. The distal tracheal region will also be examined using a fiberoptic bronchoscope introduced through the VLMA lumen prior to device removal, to assess potential blood contamination. Perioperative parameters (e.g., ventilation metrics, hemodynamic data) and postoperative recovery outcomes will be recorded and analyzed.
  Interventions: Device: Video Laryngeal Mask Airway (VLMA)
- ETT Group: Participants in this group will receive airway management using a standard endotracheal tube (ETT) inserted via direct laryngoscopy. At the end of surgery, the distal tracheal region will be examined through the endotracheal tube using a fiberoptic bronchoscope to assess the presence of blood contamination. Perioperative parameters (e.g., ventilation metrics, hemodynamic data) and postoperative recovery outcomes will be recorded and compared with those of the VLMA group.
  Interventions: Device: Endotracheal Tube (ETT)

INTERVENTIONS:
Device: Video Laryngeal Mask Airway (VLMA) — A second-generation supraglottic airway device with an integrated video camera, used for airway management in adult patients undergoing elective septoplasty. The device allows real-time visualization of the glottic inlet to identify blood infiltration or anatomical challenges. Prior to removal, a fiberoptic bronchoscope will be introduced through the device's lumen to assess the distal trachea for blood contamination. Parameters such as airway insertion time, ventilation mechanics, hemodynamic data, analgesic requirements, and postoperative recovery scores (e.g., Aldrete score, sore throat incidence) will be recorded and analyzed.
  Groups: VLMA Group
Device: Endotracheal Tube (ETT) — A standard cuffed endotracheal tube inserted using direct laryngoscopy, employed for airway management during elective septoplasty. At the end of surgery, a fiberoptic bronchoscope will be passed through the ETT to evaluate the distal trachea for blood contamination. Airway insertion time, ventilation parameters, intraoperative hemodynamics, analgesic use, and postoperative outcomes (including sore throat and recovery scores) will be documented and compared with the VLMA group to assess differences in airway safety and clinical performance.
  Groups: ETT Group

SUMMARY:
This randomized controlled trial compares a video laryngeal mask airway (VLMA) and an endotracheal tube (ETT) in adult patients undergoing elective septoplasty. The primary objective is to see which device more effectively prevents surgical blood contamination in the glottic and subglottic regions. The study also assesses perioperative hemodynamic stability, ventilation parameters, and postoperative recovery factors such as sore throat, hoarseness, and overall patient comfort. The findings aim to help determine the optimal airway device choice for nasal surgeries.

DETAILED DESCRIPTION:
This prospective, randomized controlled trial will compare the efficacy and safety of a video laryngeal mask airway (VLMA) versus a standard endotracheal tube (ETT) for airway management in adult patients (aged 18-65, ASA physical status I-II) undergoing elective septoplasty under general anesthesia.

Participants will be randomly assigned to receive either a video-assisted supraglottic airway (VLMA) or a conventional endotracheal tube (ETT). The primary objective is to evaluate whether VLMA can provide better protection against blood contamination in the glottic and subglottic regions compared to ETT. Secondary objectives include assessments of perioperative hemodynamic stability, respiratory performance, postoperative airway-related complications, and overall recovery.

All patients will undergo standardized anesthesia induction (e.g., propofol plus an opioid) and maintenance with inhalational agents and/or remifentanil infusion. Depth of anesthesia will be monitored using the bispectral index (BIS), along with standard ASA monitoring. Respiratory parameters (tidal volume, end-tidal CO₂, peak and plateau airway pressures) will be recorded throughout the procedure. Hemodynamic data (heart rate, systolic and diastolic arterial pressures) will be measured at predefined time points: pre-induction, post-airway insertion, and post-extubation.

At the end of surgery, blood contamination within the airway will be assessed at two anatomical levels:

Distal trachea: In both groups, a fiberoptic bronchoscope will be used for evaluation. In the ETT group, the bronchoscope will be inserted through the endotracheal tube before removal. In the VLMA group, the bronchoscope will be passed through the lumen of the VLMA prior to removal.

Glottis/tracheal inlet: This region will be assessed only in the VLMA group, using the device's integrated video camera to obtain a direct visual inspection before removal.

A standardized four-point scale adapted from Kaplan et al. will be used to rate the degree of blood contamination:

1. = No visible blood,
2. = Mild contamination,
3. = Moderate contamination,
4. = Severe contamination with diffuse blood.

Following airway device removal, all patients will be transferred to the post-anesthesia care unit (PACU) and monitored until achieving an acceptable Aldrete score. Postoperative airway-related symptoms-such as sore throat, hoarseness, dysphagia, and cough-will be assessed at 2, 8, 12, 24, and 48 hours. Additional data including total anesthesia duration, airway insertion time, and any adverse events (e.g., laryngospasm, bronchospasm, desaturation, or need for airway repositioning) will also be documented.

This study aims to determine whether VLMA offers advantages over ETT in terms of airway protection, intraoperative stability, and postoperative comfort in septoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II classification patients
* Patients aged 18-65 years undergoing elective septoplasty

Exclusion Criteria:

* ASA III-IV classification patients
* Patients with anticipated difficult airway
* Patients under 18 years of age
* History of gastroesophageal reflux disease (GERD) or hiatal hernia
* Body mass index (BMI) >30
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (aged 18-65 years) undergoing elective septoplasty under general anesthesia. Participants are classified as ASA I-II and are randomly assigned to the VLMA or ETT groups. Patients with anticipated difficult airway, high BMI (>30), GERD, or pregnancy are excluded
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Glottis/Trachea and Distal Trachea Blood Contamination Scores | Evaluated once at the conclusion of surgery, immediately prior to device removal (approximately 60-120 minutes after anesthesia induction).
  The presence of blood contamination will be evaluated separately at two distinct airway sites:
  Distal trachea: Both SaCoVLM and ETT groups will undergo fiberoptic bronchoscopic evaluation for blood contamination in the distal trachea immediately before removal of the airway device at the end of surgery.
  Glottis/tracheal inlet: This area will be visually assessed only in the SaCoVLM group using the integrated camera of the video laryngeal mask immediately prior to device removal at the end of surgery.
  A standardized 4-point scale will be used for both assessments:
  1. = No blood contamination
  2. = Mild amount of blood contamination (trace amounts)
  3. = Moderate amount of blood contamination
  4. = Severe amount of blood contamination

SECONDARY OUTCOMES:
Heart Rate (HR) | From preoperative baseline until arrival to the recovery unit (approximately 120 minutes).
  Heart rate (beats per minute) will be recorded at the following time points: pre-operative baseline; immediately after induction of anesthesia; at 1, 3, 5, 10, 15, and 30 minutes after airway-device insertion; and at 5 minutes after extubation.
Postoperative Sore Throat (POST Score) | Up to 48 hours postoperatively.
  he severity of postoperative sore throat (POST) will be assessed using a standardized scoring system immediately after extubation, upon arrival to the recovery room, and at 2, 8, 12, 24, and 48 hours postoperatively. The score is based on patient-reported discomfort and classified as follows: 0: No sore throat
  1. Mild discomfort (less than a common cold)
  2. Moderate discomfort (as bad as a common cold)
  3. Severe discomfort interfering with daily activities The assessment will be conducted through direct patient questioning at each designated time point.
Arterial Blood Pressure (Systolic, Diastolic, and Mean) | From preoperative baseline until arrival to the recovery unit (approximately 120 minutes).
  Systolic, diastolic, and mean arterial blood pressures (mmHg) will be recorded at the following time points: pre-operative baseline; immediately after induction of anesthesia; at 1, 3, 5, 10, 15, and 30 minutes after airway-device insertion; and at 5 minutes after extubation.
Total Remifentanil Consumption | Intraoperative
  Total remifentanil dose (mcg) administered during surgery will be compared between groups.
Airway Insertion Time | Immediately after induction of anesthesia
  The time required to successfully place the assigned airway device (VLMA or ETT), measured from the moment the device is picked up until effective ventilation is confirmed via capnography and chest rise. This outcome evaluates the ease and efficiency of airway device placement.
Intraoperative Airway Complications | From induction of anesthesia to extubation (intraoperative period)
  Incidence of intraoperative airway complications such as bronchospasm, laryngospasm, airway obstruction, or intraoperative desaturation episodes (SpO₂ <90%) will be systematically recorded.
Postoperative Dysphagia (Swallowing Difficulty) | Up to 48 hours postoperatively.
  Presence or absence of swallowing difficulty (dysphagia) will be evaluated immediately after extubation, upon arrival to the recovery room, and at 2, 8, 12, 24, and 48 hours postoperatively using direct patient questioning.
First-Attempt Success Rate of Airway Device Insertion | Immediately after induction of anesthesia.
  Comparison of the success rate of airway device insertion (VLMA or ETT) at the first attempt. Additionally, the total number of insertion attempts required for successful placement will be evaluated.
Postoperative Nausea and Vomiting (PONV) | Up to 48 hours postoperatively.
  Presence or absence of postoperative nausea and vomiting (PONV) will be assessed immediately after extubation, upon arrival to the recovery room, and at 2, 8, 12, 24, and 48 hours postoperatively using direct patient questioning.
Airway Pressure Parameters (Peak and Mean Airway Pressure) | From 1 minute to 30 minutes after airway device placement.
  Peak inspiratory pressure (PIP) will be measured and recorded at 1, 3, 5, 10, 15, and 30 minutes after airway-device insertion.
Anesthesia Duration | Intraoperative period (approximately 60-120 minutes)
  Total duration of anesthesia will be measured from the start of induction to the transfer of the patient to the recovery unit.
Surgical Duration | Intraoperative period (approximately 30-120 minutes)
  Duration of surgery will be recorded from the initial surgical incision to the completion of the final suture.
Postoperative Laryngospasm and Bronchospasm | Within 24 hours post-extubation
  The incidence of postoperative laryngospasm and bronchospasm will be assessed clinically within the first 24 hours following extubation. Laryngospasm is defined as an involuntary spasm of the vocal cords resulting in airway obstruction, while bronchospasm refers to a sudden constriction of the bronchial muscles leading to respiratory distress. These conditions will be diagnosed based on clinical signs such as stridor, increased respiratory effort, reduced airflow, and desaturation (SpO₂ <90%).

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Selcuk KUSDERCI, M.D., Study Director — Samsun University
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaplan A, Crosby GJ, Bhattacharyya N. Airway protection and the laryngeal mask airway in sinus and nasal surgery. Laryngoscope. 2004 Apr;114(4):652-5. doi: 10.1097/00005537-200404000-00010. PMID 15064618
- [Background] Karaaslan E, Akbas S, Ozkan AS, Colak C, Begec Z. A comparison of laryngeal mask airway-supreme and endotracheal tube use with respect to airway protection in patients undergoing septoplasty: a randomized, single-blind, controlled clinical trial. BMC Anesthesiol. 2021 Jan 7;21(1):5. doi: 10.1186/s12871-020-01222-4. PMID 33407130
- See also: Relevant study comparing LMA and ETT in septoplasty (Karasalan et al., BMC Anesthesiol 2021) — https://pubmed.ncbi.nlm.nih.gov/33407130/